CLINICAL TRIAL: NCT00344552
Title: Phase II Study to Evaluate Efficacy and Safety of Weekly Paclitaxel (BMS-181339)in Patients With Advanced or Recurrent Esophageal Cancer. This Study is an Extension Study for Japanese Registration Only.
Brief Title: Phase II Study of Weekly Paclitaxel (BMS-181339)in Patients With Advanced or Recurrent Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-540
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Injection solution, IV, 100mg/sqm, once weekly, 7 weeks and over
  Other Names: Taxol

SUMMARY:
The purpose of this clinical research study is to learn if BMS-181339 can shrink or slow the growth of the cancer in patients with advanced or recurrent esophageal cancer. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable disease
* Patients must have experienced on pervious chemotherapy regime
* Men and Women, with the age 20 years or older
* ECOG PS: 0-1

Exclusion Criteria:

* Patients with previous therapy with Taxanes

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate | at the end of the study
Safety | at the end of the study

SECONDARY OUTCOMES:
Response duration | at the end of the study
Time to progression (TTP) | at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- Japan (12):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kashiwa-Shi, Chiba
  - Local Institution, Sagamihara-Shi, Kanagawa
  - Local Institution, Osaka, Osaka
  - Local Institution, Ōsaka-sayama, Osaka
  - Local Institution, Suita-Shi, Osaka
  - Local Institution, Takatsuki-Shi, Osaka
  - Local Institution, Saitama, Saitama
  - Local Institution, Sunto-Gun, Shizuoka
  - Local Institution, Utsunomiya, Tochigi
  - Local Institution, Chuo-Ku, Tokyo
  - Local Institution, Toshima-Ku, Tokyo